CLINICAL TRIAL: NCT03929185
Title: Study of the Chemical Pattern Exhaled by Different Neoplasms Through Chemoresistive Sensors in Order to Identify Specific Biomarkers. Pre-clinic Evaluation
Brief Title: Analysis of Chemical Pattern Exhaled by Different Neoplasms Through Chemoresistive Nanostructured Sensors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Gabriele Anania, Professor, University Hospital of Ferrara
Other Study IDs: 170484
Record Dates: First submitted 2019-04-17; First posted 2019-04-26 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Tumor, Solid
Keywords: Volatile organic compounds; colorectal cancer; non invasive diagnostic tests; medical device
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood and tumor biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tumor affected: Patients affected by colorectal cancer who underwent to surgical resection in Sant'Anna Hospital in Cona (Ferrara)
  Interventions: Diagnostic Test: blood analysis with SCENT B1; Diagnostic Test: tissue analysis with SCENT B1
- Control: Healthy people aged 20-35 years old without risk factors for colorectal cancers who voluntarily participated to the study
  Interventions: Diagnostic Test: blood analysis with SCENT B1

INTERVENTIONS:
Diagnostic Test: blood analysis with SCENT B1 — analyze blood samples with chemoresistive sensors
  Other Names: patent number: 102015000057717
Diagnostic Test: tissue analysis with SCENT B1 — analyze tumor biopsies collected during surgery with chemoresistive sensors
  Other Names: patent number: 102015000057717
  Groups: Tumor affected

SUMMARY:
The aim of the study is to identify a pattern of chemoresistive sensors able to recognise the presence of a tumoral pathology from a health state through the analysis of Volatile Organic Compounds inside the specimen.

The chemoresistive nanostructured sensors are into an innovative patented device SCENT B1 which can analyse different specimens: blood samples, tissue biopsies, cell cultures.

In this study SCENT B1 wil be used to compare the measures of:

* tumoral and health tissues taken from different neoplasms after their surgical resection
* blood samples from healthy and tumor affected people
* pre and post- operative blood samples of tumor affected people

DETAILED DESCRIPTION:
SCENT B1 is a patented device constituted by four chemoresistive nanostructured sensors able to vary their conductance depending on chemical substances present in the environment. These sensors are extremely sensitive as they can identify substances at a concentration of tens parts per billion such as volatile organic compounds derived from tumor cells metabolism.

Every sensor answers differently from the others and the aim of the study is to find the best array of sensors able to discriminate among tumoral and healthy specimens.

Different specimens are tested: tissue biopsies and blood samples. Blood samples are collected from patients undergoing surgical resection of the neoplasm. A first blood sample is collected before the surgery and it is compared to a control sample taken from an healthy volunteer. The second blood sample is taken from the patient during a follow-up visit after the finish of any post-operative therapy. Blood samples are conserved at ambient temperature and analyzed by SCENT B1 on the same day of the collection.

Health and tumoral tissue biopsies are collected from surgical resection specimens, kept in breeding ground, cleaned from bacteria, adipose tissue and other contaminants and finally processed in SCENT B1 on the day after the collection.

The four sensors' outputs are combined in statistical analysis in order to define the threshold between health and tumor affected specimens.

ELIGIBILITY:
Inclusion Criteria:

* patients who undergo to open or laparoscopic surgery for colorectal cancer in election regimen
* patients who underwent to open or laparoscopic surgery for colorectal cancer and who have finished chemotherapy or radiotherapy yet

Exclusion Criteria:

* patients operated in emergency regimen
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People coming to Sant'Anna University Hospital of Cona, Ferrara (Italy)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-07-13 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
capability of SCENT B1 to distinguish healthy and tumoral specimens | up to 3 days after surgery for each patient
  Analysis of the difference in voltage outputs of the array of sensors when exposed to healthy and tumoral specimens. Data are statistically combined in order to find the threshold value that distinguish healthy from tumor affected conditions

SECONDARY OUTCOMES:
capability of SCENT B1 to monitor cancer recurrences | during the post-treatment follow-up visit for each patient, an average of 1 year
  comparison of SCENT B1 responses to blood samples taken from the same patient in different moments before and after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Anania, Principal Investigator — Società Italiana Chirurgia Endoscopica
Locations (1):
- Istituto di chirurgia generale 1, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No
privacy